CLINICAL TRIAL: NCT06250725
Title: Sleep Enhancement for Older Adults Living With Memory Loss And Their Care Partners
Acronym: SLEEPMATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Glenna Brewster, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00006711; 5K23AG070378-03 (NIH)
Record Dates: First submitted 2024-02-01; First posted 2024-02-09 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Sleep Disturbance; Dementia
Keywords: Persons living with dementia (PLwD); Caregivers; Cognitive Behavioral Therapy for Insomnia (CBTi)
MeSH Terms: conditions — Parasomnias; Dementia | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cognitive Behavioral Therapy for Insomnia (CBTi) (Experimental): Participant dyads will receive CBTi via videoconferencing sessions
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — The intervention protocol will include CBTi principles like stimulus control, sleep compression, relaxation, sleep hygiene, and cognitive restructuring. It will be done over 6 weeks with one session weekly via videoconference.
  Other Names: CBTi

SUMMARY:
The purpose of this study is to determine if a 6-week videoconference intervention to teach skills to improve sleep is practical, acceptable, and helpful to persons living with memory loss, cognitive impairment, and/or dementia and care partners, individually or together.

DETAILED DESCRIPTION:
Disturbed sleep is stressful to persons living with dementia (PLwD) and their caregivers. It contributes to the earlier placement of the PLwD in nursing homes and increases the risk for many psychological and cognitive health issues and poor quality of life for both the PLwD and the caregivers. Given the potential harmful side effects of medications, non-medication alternatives, such as Cognitive Behavioral Therapy for Insomnia (CBTi), may be safer to improve disturbed sleep in this population. CBTi which includes stimulus control, sleep compression, relaxation, sleep hygiene, and cognitive restructuring, is effective and has durable and sustained effects on sleep outcomes over the long term. CBTi has improved sleep disturbances in PLwD and their caregivers, separately. Since disturbed sleep in the PLwD-caregiver dyad is bidirectional and interdependent, targeting the pair as a unit for intervention has the potential to lead to improved sleep and health outcomes for both persons.

There is no current published research on CBTi when the PLwD and their caregivers receive the intervention at the same time; as a result, the research team aims to examine the 1) feasibility and 2) preliminary efficacy of 6-week CBTi intervention for community-dwelling PLwD and their caregivers who are both experiencing sleep disturbances. PLwD-caregiver dyads will participate in videoconferencing sessions. In addition, semi-structured interviews will take place to examine the acceptability and satisfaction with the intervention.

ELIGIBILITY:
Inclusion Criteria for the PLwCI:

* Diagnosis of Alzheimer's Disease and Related Dementias (ADRD), or caregiver-reported probable or possible cognitive impairment or
* Montreal Cognitive Assessment (MOCA) score between 12 and 24;
* Had ≥1 sleep problem ≥3x/week on the Neuropsychiatric Inventory (NPI)-Nighttime Behavior Subscale;
* Have an eligible caregiver;
* Be able to participate in the intervention sessions

Inclusion Criteria for Caregivers:

* ≥18 years old, co-residing with persons living with cognitive impairment (PLwCI);
* Regularly assist the care recipient with ≥1 of 7 basic activities of daily living or
* ≥1 of 7 Instrumental Activities of Daily Living for the past 6 months;
* Have difficulty falling asleep or difficulty staying asleep for the last three months or
* Have a Pittsburgh Sleep Quality Index (PSQI) of 5 or greater

Exclusion Criteria:

* PLwCI: Moderate to severe cognitive impairment
* Individuals who are not yet adults
* Pregnant women
* Prisoners
* Individuals who are not able to clearly understand English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change in insomnia | Baseline, 1-week post-intervention, and 3 months post-intervention
  Insomnia will be measured using the Insomnia Severity Index. The insomnia severity index ahs seven questions. The seven answers are added up to get a total score.
  Total score categories:
  0-7= No clinically significant insomnia 8-14= Subthreshold insomnia 15-21= Clinical insomnia (moderate severity) 22-28= Clinical insomnia (Severe)
Change in Sleep Efficiency | Baseline, 1-week post-intervention, and 3 months post-intervention
  Sleep Efficiency will be measured using sleep diaries and actigraphy. Actigraphy watches monitor sleep-wake cycles by recording activity patterns continuously. Participants will also complete a diary each morning that asks about their sleep-wake patterns.
Change in in Sleep Onset Latency | Baseline, 1-week post-intervention, and 3 months post-intervention
  Sleep onset latency will be measured using sleep diaries and actigraphy. Actigraphy watches monitor sleep-wake cycles by recording activity patterns continuously. Participants will also complete a diary each morning that asks about their sleep-wake patterns.
Change in Wake After Sleep Onset | Baseline, 1-week post-intervention, and 3 months post-intervention
  Wake after sleep onset will be measured using sleep diaries and actigraphy. Actigraphy watches monitor sleep-wake cycles by recording activity patterns continuously. Participants will also complete a diary each morning that asks about their sleep-wake patterns.
Adherence with Study Interventions (feasibility) | weekly during the intervention period up to 3 months post-intervention
  Feasibility of the interventions will be assessed with rates of adherence to the study components throughout the study participation.
Satisfaction with intervention components | 1 week post-intervention
  Satisfaction with the intervention components will be assessed with the study satisfaction measure questionnaire that has 16 questions type that uses an agree, disagree scale as a range of answer options that go from strongly agree to strongly disagree.

SECONDARY OUTCOMES:
Change in depression | Baseline, 1-week post-intervention, and 3 months post-intervention
  Depression will be measured using the Center for Epidemiologic Studies Depression scale. The Center for Epidemiologic Studies Depression scale has 20 questions. The 20 answers are added up to get a total score between 0 and 60.
  Total score categories:
  16 or greater = Clinically significant depressive symptoms
Change in the Quality of Life | Baseline, 1-week post-intervention, and 3 months post-intervention
  Quality of Life will be measured using the research and development (RAND) Medical Outcomes short form (SF)-36. The insomnia severity index has 36 questions which have subscales that total 100. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.

CONTACTS AND LOCATIONS:
Overall Officials: Glenna Brewster, PhD, RN, FNP, Principal Investigator — Emory University
Locations (1):
- Emory Healthcare System, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The research team will share the participants' research identification with instrument responses.
Supporting Information: Study Protocol
Time Frame: Starting 01/01/2028
Access Criteria: Requests can be sent to the PI with a document that includes the background and research questions to conduct secondary data analyses.